CLINICAL TRIAL: NCT00005424
Title: Prospective Analysis of the Effect of Widowhood on CVD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4342; R03HL049043 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine the effect of widowhood on cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Widowed persons have been found to have higher mortality rates than married persons in both cross-sectional and longitudinal studies. In many of these studies, excess mortality has been attributed to deaths from cardiovascular disease. Despite these consistent findings, the lack of detailed data collected prior to widowhood has hampered our ability to understand the mechanisms to explain this effect. Furthermore, an understanding of the mechanisms underlying this effect might help elucidate the apparent gender differences in mortality following widowhood.

DESIGN NARRATIVE:

The study took advantage of the data collected as part of the Framingham Study to investigate the effect of widowhood on cardiovascular disease. The Framingham dataset has extensive clinical data related to cardiovascular disease, as well as to health behaviors. These longitudinal data provided the opportunity to prospectively characterize the health of widows prior to and following the loss of a spouse in much greater detail than previously possible. The analyses used a prospective design in which those men and women who had a spouse die during the course of the study (N=626) were compared to men and women who remained married (N=2044). These analyses also provided the opportunity to examine reasons for the beneficial effect found of remarriage. The study addressed the following questions: 1. Can the increased risk of mortality from cardiovascular disease often found following widowhood be explained by pre-widowhood health status? 2. Can increased mortality following widowhood be explained by changes in health behaviors related to cardiovascular disease risk. 3. What pre-widowhood risk factors place the widowed at greater risk for cardiovascular disease morbidity and/or mortality following the death of a spouse? 4. Can pre-widowhood risk factors or post-widowhood behavior change account for gender differences in mortality following widowhood?

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1996-02 (Actual)